CLINICAL TRIAL: NCT03724149
Title: Open-Labeled Trial Of Direct-acting Antiviral Treatment Of Hepatitis C-Negative Patients Who Receive Lung Transplants From Hepatitis C-Positive Donors
Brief Title: Transplanting Hepatitis C Lungs Into Negative Lung Recipients
Acronym: SHELTER
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 829397
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Results first posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Lung Diseases
Keywords: Lung Disease
MeSH Terms: conditions — Lung Diseases | interventions — elbasvir-grazoprevir drug combination; sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Direct-acting antiviral treatment for HCV (Experimental)
  Interventions: Drug: Zepatier; Drug: Epclusa

INTERVENTIONS:
Drug: Zepatier — Zepatier (grazoprevir 100mg and elbasvir 50 mg once daily) is taken by mouth for 12 weeks unless a genetic variation is detected. In this case treatment with Zepatier will be extended to 16 weeks. Study subjects with treatment failure will be provided open-label Zepatier + sofosbuvir (sovaldi) 400mg + Ribavirin (generic), renally dosed based on creatinine clearance per the manufacturer guidelines.
Drug: Epclusa — Epclusa (sofosbuvir 400mg and velpatasvir 100mg once daily) is taken by mouth for 12 weeks. Study subjects with treatment failure will be provided an alternative DAA + sofosbuvir (sovaldi) 400mg + Ribavirin (generic), renally dosed based on creatinine clearance per the manufacturer guidelines.

SUMMARY:
This study is being conducted to determine safety and effectiveness of transplanting lungs from Hepatitis C-positive donors into Hepatitis C-negative patients on the lung transplant waitlist, who will then be treated with appropriate direct-acting antiviral (DAA) after transplantation.

DETAILED DESCRIPTION:
Open-labelled pilot clinical trial of Zepatier (Grazoprevir + Elbasvir), Epclusa (Sofosbuvir + Velpatasvir), or another appropriate DAA in at least 10 HCV-negative subjects receiving a lung transplant from a hepatitis C (HCV)-positive donor. Eligible subjects will receive a lung transplant from a deceased-donor, and then will receive treatment after lung transplantation when infection with HCV is confirmed in these lung transplant recipients. Treatment will be complete after 12 weeks for most subjects.

ELIGIBILITY:
Subject Selection Criteria

Inclusion Criteria:

* 18-67 years of age
* Obtained agreement for participation from the lung transplant team
* No evident contraindication to lung transplantation other than the underlying lung disorder
* Able to travel to the University of Pennsylvania for routine post-transplant visits and study visits for a minimum of 12 months after transplantation
* No active illicit substance abuse
* Women must agree to use birth control in accordance with Mycophenolate Risk Evaluation and Mitigation Strategy (REMS) following transplant due to the increased risk of birth defects and/or miscarriage
* Both men and women must agree to use at least one barrier method of birth control or remain abstinent following transplant due to risk of HCV transmission
* Inclusion criteria for treatment (not for entry as study patient) will include any detectable HCV RNA by week 4 post-lung transplantation
* Able to provide informed consent

Exclusion Criteria:

* Hepatocellular carcinoma
* HIV positive
* HCV RNA positive
* Hepatitis B surface antigen and/or DNA positive
* Any chronic liver disease (excluding non-alcoholic fatty liver disease (NAFLD)) that is occurring in the setting of persistently elevated liver enzymes (patients with Alpha-1-antitrypsin lung disease without hepatic involvement are eligible)
* Significant fibrosis (≥F2 on the Fibroscan)-for patients with cystic fibrosis, the cutoff will be 11kPa (cutoff for F2 for patients with chronic cholestatic liver disease), whereas for all other patients the cutoff will be 8kPa (the cutoff for fatty liver disease used in the THINKER study).
* Pregnant or nursing (lactating) women
* Known allergy or intolerance to tacrolimus that would require post-transplant administration of cyclosporine, rather than tacrolimus given the drug-drug interaction between cyclosporine and Zepatier/Epclusa
* Pre-transplant treatment with amiodarone given the drug-drug interaction between amiodarone and Epclusa
* Waitlisted for a multi-organ transplant
* Patients with underlying liver disease with or without liver cirrhosis
* Patients with cystic fibrosis who have underlying liver disease
* Re-transplant candidate
* Use of ECMO or mechanical ventilation as a bridge to lung transplantation
* Inability to provide study consent
* Chronic kidney disease with GFR<50 ml/min/1.73 m^2

Relative contraindications for study subjects that will be reviewed on a case-by-case basis by the Lung Transplant Selection Committee and the Principal Investigators:

* Evidence of end organ damage due to diabetes (e.g. retinopathy, nephropathy, ulcerations) and /or brittle diabetes mellitus (e.g. history of diabetic ketoacidosis) and/or uncontrolled diabetes as evidence by a HgbA1C of 7.5-8.5.
* Hematologic: Significant coagulation abnormalities, and/or bleeding diatheses.
* Active or recent solid or liquid malignancy in the past 5 years (apart from select skin malignancies).
* Patient refusal to receive blood products or transfusions during lung transplant surgery.
* Psychosocial: Profound neurocognitive impairment with absence of social support.
* Active mental illness or psychosocial instability
* Inadequate insurance and/or financial support for post-transplant care.
* Evidence of drug, tobacco or alcohol abuse within the past six months and failure to satisfy recommended therapy/services/parameters as indicated by social work staff and/or consult team.
* History of chronic non-adherence to medical recommendations and/or medications
* PRA >10%.
* Severe malnutrition, BMI <18
* Major chronic disabling comorbidity (e.g. lupus, severe arthritis, neurologic diseases, previous stroke with profound residual).
* Symptomatic or severe vascular disease (History of CABG, Aorta-femoral surgery)

Donor Organ Selection Criteria

Broad goal: To include donors with confirmed HCV expected to have acceptable post-transplant graft outcomes based on large retrospective lung transplant studies.

Inclusion criteria for donors:

* Detectable HCV RNA
* Age ≤55 years
* PaO2/FiO2 ≥300 on FiO2 = 100% and PEEP=5
* Cigarette use history ≤20 pack years
* No evidence of cirrhosis
* No prior treatment of HCV with a DAA-based therapy
* Can be isolated hepatitis B Core IgG positive, but cannot have a detectable HBV Core IgM, HBSAg, and/or HBV DNA (positive HBV NAT test)

Donor Exclusion Criteria:

* Donation after circulatory death determination (DCDD)
* HIV positive

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Reese, MD, MSCE, Study Director — Perelman School of Medicine at the University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Direct-acting Antiviral Treatment for HCV
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Direct-acting Antiviral Treatment for HCV
Number analyzed (Participants) | 10
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Age | 57 [44 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Blood type [Count of Participants; unit: Participants]
  A | 2
  O | 8

OUTCOME MEASURES:

1. Primary Outcome: Subject Sustained Virologic Response (SVR-12) at 12-weeks Post-treatment
Description: The primary outcome measure is Sustained Virologic Response (SVR) rate at 12 weeks (number of subjects with SVR; negative HCV RNA after completing therapy) / (number of subjects treated post-lung transplantation).
  SVR will be based on the standard definition of SVR-12, defined as an undetectable HCV RNA in a subject's serum 12 weeks after completing treatment for HCV (12 weeks after the subject takes the last dose of Zepatier, Epclusa, or another appropriate antiviral treatment).
Time Frame: Baseline to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Direct-acting Antiviral Treatment for HCV
Number analyzed (Participants) | 10
Participants | 10

2. Primary Outcome: Major Adverse Events Attributable to HCV Therapy in Post-lung Transplant Patients Post-lung Transplant Patients
Time Frame: Baseline to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Direct-acting Antiviral Treatment for HCV
Number analyzed (Participants) | 10
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 year post-transplant
Arm/Group | Direct-acting Antiviral Treatment for HCV
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Direct-acting Antiviral Treatment for HCV (N=10)
Severe acute kidney injury (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT03724149/Prot_SAP_001.pdf